CLINICAL TRIAL: NCT02901964
Title: Effect of Strengthening the Hip Abductor in Patients With Knee Osteoarthritis: Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Ceara (Other)
Responsible Party: Principal Investigator, Gabriel Peixoto Leão Almeida, Professor, Universidade Federal do Ceara
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Doutorado
Record Dates: First submitted 2016-09-05; First posted 2016-09-15 (Estimated); Last update posted 2018-11-02 (Actual); Status verified 2018-10

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group Hip Abductor Exercise (Experimental): 12 treatments sessions at 6 weeks: Heating, lower limb stretching, tibiofemoral and patellofemoral mobilization, strengthening the quadriceps, hamstrings, triceps sural and hip abductors.
  Interventions: Other: Hip Abductor Exercise
- Group Hip Aductor Exercise (Active Comparator): 12 treatments sessions at 6 weeks: Heating, lower limb stretching, tibiofemoral and patellofemoral mobilization, strengthening the quadriceps, hamstrings, triceps sural and hip aductors.
  Interventions: Other: Hip Aductor Exercise

INTERVENTIONS:
Other: Hip Abductor Exercise — 12 treatments sessions at 6 weeks: Heating, lower limb stretching, tibiofemoral and patellofemoral mobilization, strengthening the quadriceps, hamstrings, triceps sural and hip abductors.
  Arms: Group Hip Abductor Exercise
Other: Hip Aductor Exercise — 12 treatments sessions at 6 weeks: Heating, lower limb stretching, tibiofemoral and patellofemoral mobilization, strengthening the quadriceps, hamstrings, triceps sural and hip aductors.
  Arms: Group Hip Aductor Exercise

SUMMARY:
Osteoarthritis (OA) is a prevalent disease associated with significant morbidity and is one of the most common causes of joint pain. Characterized by their chronicity, slow and progressive evolution. The overall prevalence of symptomatic knee osteoarthritis is estimated at 3.8%, with peak prevalence in the population with an average age of 50 years. The main objectives of interventions in patients with knee OA are reduced pain and improved functional capacity and exercises are widely recommended. The literature shows a lack of clinical trials verifying the effect of strengthening the hip muscles in patients with knee osteoarthritis. Thus, the aim of this study is to assess the effect of strengthening the hip abductor muscles versus hip adductor muscles in patients with symptomatic OA of the knee.

DETAILED DESCRIPTION:
The physical therapy sessions will average duration of one hour, often twice a week for six weeks. The exercise intensity will be monitored by the physiotherapist as determined by the participant's ability to complete 10 repetitions for a particular exercise and its difficulty of execution perceived by the modified Borg scale (CR-10). The exercises are performed with load between 60-80% of their capacity, the load will be increased from 2 to 10% when the patient can perform 14 full repetitions in the last series (76). It will be set to 30 seconds of rest between reps and 2 minutes between sets of exercise.

Both groups will perform prior heating exercises exercise bike for 10 minutes with moderate intensity with the Borg scale. Then there will be two stretches repetitions held for 30 seconds of muscle groups: hamstrings, quadriceps, abductors, adductors and gastrocnemius. Manual therapy for patellofemoral and tibiofemoral joint will be held after the completion of stretching. Recent clinical guidelines on knee OA strongly recommend the use of strengthening exercises of the lower limbs, both in closed kinetic chain and open. Thus, they will be performed strengthening exercises in extension and knee flexion in open kinetic chain, squat up and down a step and exercises to sural triceps. For symptom control during exercise in CKC will be used the numeric scale of pain before and after its execution.

The GABQ add the hip abduction exercises in lateral decubitus, exercise "Clam" and pelvic elevation. Studies prior point out that these exercises are among those with higher electromyographic activity of the gluteus medius muscle.

The GADQ add the adduction exercises hip in lateral recumbency, bilateral adduction with a ball between the legs and functional diagonal leg.

The exercises will be carried out to load 60-80% of 1 repetition maximum 8-12 reps, 1-3 sets and 2-3 times a week. All exercises are performed without worsening pain and intensity of exercise will be controlled according to the perceived exertion scale of Borg.

ELIGIBILITY:
Inclusion Criteria:

* OA knee radiograph grades 2 - 4 according to the Kellgren-Lawrence scale;
* Reporting knee pain with minimum intensity of 3 on Numerical Pain Scale;
* Complaints of pain and functional reduction in the last three months;
* Meet at least one of the American College of Rheumatology classification criteria;
* Deambulation independent;
* Absence of prostheses or orthoses
* Predominant pain in the medial aspect of the knee.

Exclusion Criteria:

* Contraindications for physical exercises evaluated by the Physical Activity Readiness Questionnaire (PAR-Q);
* Diabetes type I or decompensated;
* Hypertension decompensated;
* Cardiac pacemaker;
* Cancer History
* Neurological deficits (sensory or motor)
* Body mass index above 40 kg / m2
* Hip symptomatic osteoarthriti
* Orthopedic surgery of the lower limbs
* Systemic inflammatory disease
* Can not walk.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2016-09; Primary Completion 2018-05 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Scale | Six weeks
  Pain was assessed by use of an 11-point Numeric Pain Scale, where 0 corresponded to no pain and 10 corresponded to worst imaginable pain.
Pain and Function subscale - Knee Injury and Osteoarthritis Outcome Score | Six weeks
  Pain and Function subscale - KOOS was assessed, where 0 corresponded to no pain and normal function and 100 corresponded to worst pain and function.

SECONDARY OUTCOMES:
Others subscales - Knee Injury and Osteoarthritis Outcome Score | Six weeks
30 s Chair Stand Test | Six weeks
Timed Up & Go Test | Six weeks
Global Perceived Effect Scale | Six weeks
Numeric Pain Scale | Six months
Knee Injury and Osteoarthritis Outcome Score | Six months
Global Perceived Effect Scale | Six months

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Peixoto Leão Almeida, PhD student, Principal Investigator — Federal University of Ceará (UFC), Brazil.
Locations (1):
- Federal University of Ceara, Fortaleza, Ceará, Brazil

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared.